CLINICAL TRIAL: NCT01875237
Title: A Phase 1/2 Trial Evaluating Treatment of Emergent Graft Versus Host Disease (GvHD) With AP1903 After Planned Donor Infusions (DLIs) of T-cells Genetically Modified With the iCasp9 Suicide Gene in Patients With Hematologic Malignancies
Brief Title: Donor Lymphocyte Infusion (DLI) of T-cells Genetically Modified With iCasp9 Suicide Gene
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0501; NCI-2013-01666 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Leukemia; Myeloma; Myeloproliferative Diseases
Keywords: Leukemia; Myeloma; Myeloproliferative Diseases; Myelodysplastic syndrome; MDS; Lymphoma; Hodgkin disease; Multiple myeloma; MM; Transplant donor; T-cells; G-versus-host disease; GvHD; G-CSF; Filgrastim; Neupogen; Fludarabine; Fludarabine phosphate; Fludara; Melphalan; Alkeran; Alemtuzumab; CAMPATH-1H; Campath; Tacrolimus; Prograf; Mini-methotrexate; AP 1903; Methylprednisolone; Depo-Medrol; Medrol; Solu-Medrol; Stem cell infusion; Donor lymphocyte infusion; DLI; Questionnaire; Survey
MeSH Terms: conditions — Leukemia; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Lymphoma; Hodgkin Disease; Multiple Myeloma | interventions — fludarabine; fludarabine phosphate; Melphalan; Alemtuzumab; Tacrolimus; Granulocyte Colony-Stimulating Factor; Filgrastim; AP 1903 reagent; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stem Cell Transplant + Modified T-Cells + Chemotherapy (Experimental): The first component is stem cell transplant. Goal is to administer more than 3 x 106 CD34+ cells/kg of peripheral blood progenitor cells (PBPC). The second component is the planned DLI infusion. iCasp9 (BPZ-1001)-Modified T-cells) of 3 X 10^6/kg in 100 ml infused over approximately a one hour period between Day + 56 to Day +64. The transplant day is referred to as day zero (D0), treatment plan activities prior or after D0 are denoted as day minus (D-) or day plus (D+). Patients receive standard reduced intensity regimen using fludarabine, melphalan, and alemtuzumab to achieve engraftment with a low risk of GVHD. At approximately 60 days post transplant patients who are alive and without GVHD, receive DLI to enhance graft-vs.-malignancy and immune reconstitution.
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Alemtuzumab; Procedure: Stem Cell infusion; Drug: Tacrolimus; Drug: Mini Methotrexate; Drug: G-CSF; Procedure: Donor Lymphocyte Infusion (DLI); Drug: AP1903; Drug: Methylprednisolone; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Fludarabine — 40 mg/m2 by vein on Days -6 to -3.
  Other Names: Fludarabine phosphate; Fludara
Drug: Melphalan — 140 mg/m2 by vein on Day -2.
  Other Names: Alkeran
Drug: Alemtuzumab — 50 mg by vein on Day -1.
  Other Names: CAMPATH-1H; Campath
Procedure: Stem Cell infusion — Stem cell infusion on Day 0. Goal is to administer more than 3 x 10^6 CD34+ cells/kg of peripheral blood progenitor cells (PBPC).
Drug: Tacrolimus — Starting dose of 0.015 mg/kg (ideal body weight) as a 24 hour continuous infusion daily adjusted to achieve a therapeutic level of 5-15 ng/ml (target is 10 ng/ml) between Day +1 and Day +45. Tacrolimus is changed to oral dosing when tolerated. Tacrolimus tapering should start on approximately Day +35 with the intention for the patient to be completely off the drug by approximately Day +45.
  Other Names: Prograf
Drug: Mini Methotrexate — 5 mg/m2 by vein on Days +1, +3, +6.
Drug: G-CSF — 5 mcg/kg/day subcutaneously beginning on Day +7, and continuing until the absolute neutrophil count (ANC) is > 500 x 10/L for 3 consecutive days.
  Other Names: Filgrastim; Neupogen
Procedure: Donor Lymphocyte Infusion (DLI) — iCasp9 (BPZ-1001)-Modified T-cells) of 3 X 10^6/kg in 100 ml infused over approximately a one hour period between Day + 56 to Day +64.
Drug: AP1903 — 0.4 mg/kg as a 2 hour infusion for patients that present with a clinical diagnosis of grade I GvHD. For patients with a clinical diagnosis of grade > 2 GvHD, a single dose of AP1903 0.4 mg/kg as a 2 hour infusion will be administered. Patients who fail to achieve a complete response within 72 hours of an initial dose of AP1903, or within 48 hours of a second dose of AP1903, will be maintained on this dose for no less than 7 days. Patients who experience a partial response within 72 hours may receive a second dose of AP1903. Patients whose GvHD is progressing after 7 days, have no response by 14 days, or are not in a complete response at day 28 can receive secondary therapy.
Drug: Methylprednisolone — 1.6 mg/kg per day by vein divided in 2 to 3 daily doses. Patients whose GvHD resolves as defined by a complete response within 72 hours, would have steroids stopped immediately. Patients who fail to achieve a complete response within 72 hours of an initial dose of AP1903, or within 48 hours of a second dose of AP1903, will be maintained on this dose for no less than 7 days. Steroids can then be tapered as tolerated to no less than 0.6 mg/kg per day at day 28.
  Other Names: Depo-Medrol; Medrol; Solu-Medrol
Behavioral: Questionnaire — Completion of a quality of life questionnaire that will take 10-15 minutes between Days + 28 and + 56, about twice a week until about 2 months after the T-cell infusion, and then 6 and 12 months after the stem cell transplant.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if giving genetically changed immune cells, called T-cells, after chemotherapy will improve the response to a stem cell transplant. The safety of this treatment will also be studied.

The process of changing the DNA (the genetic material in cells) of these T-cells is called "gene transfer." Researchers want to learn if these genetically-changed T-cells are effective in attacking cancer cells in patients with leukemia, MDS, lymphoma, Hodgkin disease, or MM, after they have received an allogeneic stem cell transplant.

The chemotherapy you will be given on study is fludarabine, melphalan, and alemtuzumab. These drugs are designed to stop the growth of cancer cells, which may cause the cancer cells to die. This chemotherapy is also designed to block your body's ability to reject the donor's stem cells.

Researchers also want to learn if giving AP1903 will help the symptoms of graft-versus-host disease (GvHD) that may occur after the T-cell infusion. GvHD occurs when donor cells attack the cells of the person receiving the stem cell transplant.

DETAILED DESCRIPTION:
Gene Transfer:

Gene transfer involves drawing blood from a transplant donor, and then separating out the T-cells using a machine. Researchers then perform a gene transfer to change the T-cells' DNA, and then inject the changed T-cells into the body of the patient receiving the transplant.

Study Drug Administration:

You will receive fludarabine, melphalan, and alemtuzumab to kill cancer cells and help prevent your body from rejecting the stem cells. The day you receive the stem cells is called Day 0. The days before you receive your stem cells are called minus days. The days after you receive the stem cells are called plus days.

On Day -7, you will be admitted to the hospital and given fluids by vein to hydrate you.

On Days -6 through -3, you will receive fludarabine by vein over 1 hour each day.

On Day -2, you will receive melphalan by vein over 30 minutes.

On Day -1, you will receive alemtuzumab by vein over 2 hours.

On Day 0, you will receive the stem cell transplant as a cell infusion by vein.

After the transplant, you will receive tacrolimus and methotrexate. At first, you will receive tacrolimus as a continuous (nonstop) infusion until you are able to take it by mouth. You will then take tacrolimus by mouth 2 times a day for about 3 weeks and then your doctor will tell you how to taper it off (gradually stop taking it). On Days +1, +3, +6, and +11, you will receive methotrexate by vein over 30 minutes.

You will receive filgrastim as an injection under the skin 1 time a day, starting 1 week after the transplant, until your blood cell levels return to normal. Filgrastim is designed to help with the growth of white blood cells.

Between Day +56 and +64, if you are in stable medical condition and have not developed GvHD, you will receive a donor lymphocyte infusion containing genetically modified T-cells by vein over 10-30 minutes. You will receive Benadryl (diphenhydramine) by vein over 15 minutes and Tylenol by mouth before the infusion to lower the risk of an allergic reaction.

If your doctor thinks it is needed due to medical problems, the T-cell infusion may be postponed for up to 6 months after the transplant.

If you develop symptoms of GvHD after the T-cell infusion, you must return to the clinic within 72 hours. Most cases of GVHD occur within 60 days of the T-cell infusion. If you have GvHD, you will receive AP1903 by vein and possibly steroids by mouth or by vein. If your doctor thinks it is needed, you may receive one more dose of AP1903 by vein 24-72 hours after the first dose.

If GvHD returns after the first treatment and your doctor thinks it is needed, you may receive AP1903 by vein and steroids by mouth or by vein.

Blood (about 2 tablespoons each time) will be drawn about 3 hours before you receive AP1903, about 2 hours after the AP1903 infusion, and then about 24 hours after the AP1903 infusion to check the level of genetically modified T-cells.

You will then come to the clinic every day for the next 3 days and for an additional 3 days after a second dose of AP1903, if given. In addition, you will come to the clinic on about Days +7, +14, +28, +42 and +56 after receiving AP1903. If your symptoms do not improve after receiving AP1903, you will be given standard drugs for GvHD.

Study Tests:

After the stem cell transplant but before the T-cell infusion, you will have the following tests and procedures to find out if you will be eligible for the T-cell infusion:

* You will have a physical exam.
* You will be checked for possible reactions to treatment, including GvHD.
* Blood (about 4 tablespoons) will be drawn for routine tests, to check your liver and kidney function, for chimerism studies (determination of donor or recipient cells), and to check for cytomegalovirus (CMV).
* If your doctor thinks it is needed, you will have a bone marrow aspiration and biopsy performed to check the status of the disease. To collect a bone marrow aspiration/biopsy, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.

About twice a week until about 2 months after the T-cell infusion, and then 6 and 12 months after the stem cell transplant:

* You will have a physical exam, including measurement of your height, weight and vital signs.
* Your medical history will be recorded.
* You will have be checked for possible reactions to your treatment, including GvHD.
* Blood (about 4 tablespoons) will be drawn for routine tests, to check your liver and kidney function, and to check for CMV and other infections. Part of the blood may be used for chimerism studies, if your doctor thinks it is needed.
* If your doctor thinks it is needed, you may have a bone marrow aspiration and biopsy performed to check the status of the disease and for chimerism studies.

If your doctor thinks it is needed, some tests and procedures may be repeated more frequently or at different time points during the study.

Immune System and T-cell Level Tests:

If possible, blood (about 3 tablespoons) will be drawn to check the status of the disease and your immune system function:

* 4 hours after the T-cell infusion,
* once a week for 1 month after the T-cell infusion,
* and then at 6 weeks and then about 2, 3, 6, 9, and 12 months after the T-cell infusion. °Part of the blood sample will be used to check for HAMA at 3 months after the T-cell infusion.

Part of the blood drawn will be tested to check the level and function of the infused T-cells. At 3 months after the T-cell infusion, blood (about 1 teaspoon) will be drawn to check for HAMA.

Questionnaires:

You will complete a quality of life questionnaire that will take about 5-10 minutes each time:

* When you enroll on this study
* At the time of the T-cell infusion
* If you develop symptoms of GvHD after the T-cell infusion and receive AP1903, you will complete the questionnaire before you receive AP1903, and then about 7 and 14 days after you receive AP1903.
* If you do not develop symptoms of GvHD, you will complete a questionnaire about 1 month after the T-cell infusion.

Length of Treatment:

You will be off study after your 1-year follow-up visit. You will be taken off study early if:

* not enough donor cells could be collected
* you were not eligible to receive the T-cell infusion
* you have graft failure (the donor cells did not "take")
* the disease comes back and needs another treatment
* you are unable to keep appointments
* you did not return to the clinic within 72 hours of having symptoms of GvHD
* your study doctor thinks it is in your best interest

If you are taken off study, you will receive standard of care treatment.

Long-Term Follow-Up:

For safety reasons, the U.S. Food and Drug Administration (FDA) requires that patients who receive infusions of stem cells treated with a gene transfer procedure must have long-term follow-up yearly for at least 15 years after receiving the gene transfer.

You will have blood tests performed to check to make sure you do not have a type of infection called the replication-competent retrovirus (RCR). For this test, blood (up to 4 teaspoons each time) will drawn about 1, 3, and 6 months after the T-cell infusion, then once every 6 months for 5 years, and then once a year after that for 10 years.

If the RCR test results during the first year after the T-cell infusion show that you do not have the RCR infection, the rest of your leftover blood samples (left over from RCR testing in Years 2-15) will be stored at Bellicum for safety reasons. This is so researchers can study any changes in your blood (related to RCR) that may arise in Years 2-15.

You will be asked to sign a separate consent form for a long-term follow-up study, Protocol 2006-0676. If for any reason you are unable to receive the genetically modified cells, you will not be enrolled on the long-term follow-up study.

This is an investigational study. The gene transfer or infusion with genetically-changed T-cells and the drug, AP1903, are not FDA approved or commercially available for use in this type of disease. They are currently being used for research purposes only. Fludarabine, melphalan, and alemtuzumab are commercially available and FDA approved.

Up to 35 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years and </= 65 years.
2. One of the following: a. Acute leukemia past first remission, in first or subsequent relapse, in second or greater remission. Patients in first remission should have with intermediate or high cytogenetic risk factors or flt3 mutation. Patients with relapsed disease. Patients with primary induction failure or relapse are eligible if they have < 10% bone marrow blasts, and no circulating blasts. b. Myelodysplastic syndrome with intermediate or high risk IPSS score, or treatment related MDS. c. CML resistant to tyrosine kinase treatment in a first or subsequent chronic phase or after transformation to accelerated phase or blast crisis.
3. 2 (continued): d. CLL, Lymphoma or Hodgkin's disease which has failed to achieve remission or recurred following initial chemotherapy. Patients must have at least a PR to salvage therapy, or low bulk untreated relapse (< 2 cm largest mass). e. Multiple myeloma which has relapsed or progressed and has achieved a partial response to salvage chemotherapy.
4. Patients must have one of the following donor types identified who are willing to donate peripheral blood: a. Related donor, 8/8 HLA-matched for HLA-A, -B, C and DR matched or, b. Matched Unrelated Donor (MUD), 8/8 HLA-matched for HLA A, B, C and DRB1 using allele level typing.
5. Performance score of at least 80% by Karnofsky.
6. Adequate major organ system function as demonstrated by: a. Creatinine < 1.8 mg/dl (or creatinine clearance > 40 ml/min) b. Bilirubin < 1.5 mg/dl except for Gilbert's disease c. ALT < 300 IU/ml d. Left ventricular ejection fraction equal or greater than 40%. e. Pulmonary function test (PFT) demonstrating a diffusion capacity of least 50% predicted, corrected for hemoglobin.
7. Patient or patient's legal representative, able to sign informed consent.
8. Patient or patient's legal representative, parent(s) or guardian able to provide written informed consent for the long-term follow-up gene therapy study 2006-0676.
9. The patient will need to be available for evaluation within 72 hours of symptoms of GVHD, occurring within 60 days of the planned donor lymphocyte infusion.

Exclusion Criteria:

1. Uncontrolled active infection.
2. Positive Beta HCG test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization.
3. Women of child bearing potential not willing to use an effective contraceptive measure while on study.
4. Men not willing to use an effective contraception method while on study.
5. Known sensitivity to any of the products that will be administered during the study.
6. HIV seropositive.
7. Prior allogeneic transplant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-12-27 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patient with hematologic malignancies receiving allogeneic hematopoietic transplants.
Pre-assignment Details: patients who do not have GVHD on day 42 receive genetically modified donor lymphocytes with suicide gene to be activated by drug AP1903 if GVHD occurs.
Groups:
- Transplant Only: Patients who did not move forward to DLI
- Transplat Plus DLI: Proceeded to DLI per protocol
Period: Overall Study
Arm/Group | Transplant Only | Transplat Plus DLI
Started | 2 | 1
Completed | 0 | 1
Not Completed | 2 | 0
Not completed — GVDH before DLI | 1 | 0
Not completed — DLI cells could not be produced | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transplant Only | Transplat Plus DLI | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Safety of Donor Lymphocyte Infusion Followed by Dimerizer Drug, AP1903 by Number of Participants With Adverse Events.
Description: To evaluate the safety of the infusion of inducible caspase 9 (BPZ-1001) modified T-cells followed by dimerizer drug, AP1903. Safety evaluated by number of participants with Adverse events.
Time Frame: up to 3.5 years
Population: Participant who received Donor Lymphocyte infusion and AP 1903
Measure: Count of Participants; unit: Participants
Groups:
- Transplant Only: Participants who did not move forward to DLI
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

2. Secondary Outcome: Number of Participants Assessed Post Donor Lymphocyte Infusion (DLI): Disease-free Survival & Non-relapse Mortality, Chimerism and GVHD.
Description: Participants to assess at 6 months post donor lymphocyte infusion (DLI): disease-free survival & non-relapse mortality, chimerism and GVHD
Time Frame: 6 months
Population: Transplant only participants did not receive DLI.
Measure: Count of Participants; unit: Participants
Groups:
- Transplat Plus DLI: Proceeded to DLI per protocol and developed GVHD
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 1
Participants
  disease-free survivaI | 0 | 1
  chimerism post DLI | 0 | 1
  GVHD post DLI | 0 | 1
  non-relapse mortality | 0 | 0

3. Secondary Outcome: To Assess the Incidence of Epstein-Barr Virus -PTLD or EBV Reactivation Requiring Therapy Post DLI.
Description: To assess the incidence of Epstein-Barr virus (EBV)-associated lymphoproliferative disorder or EBV reactivation requiring therapy post DLI.
Time Frame: 1 year
Population: all patients who received DLI
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

4. Secondary Outcome: To Assess the Proportion of Patients Developing Grade I-IV Acute GvHD
Description: To assess the proportion of patients developing grade I-IV acute GvHD by Day 28, 56, and 180 post DLI.
Time Frame: Day 28, 56, and 180 post DLI.
Population: all patients who received DLI
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 1
Participants
  Day 28 | 0 | 1
  Day 56 | 0 | 1
  Day 180 | 0 | 0

5. Secondary Outcome: To Assess the Proportions of GvHD Response Post-administration of AP1903.
Description: To assess the proportions of GvHD complete response (CR), partial response (PR), mixed response, no response, and progression among surviving patients at Day 3, 7, 14, 28, and 56 post-administration of AP1903.
Time Frame: Day 3, 7, 14, 28, and 56 post-administration of AP1903
Population: Patient who received DLI
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 1
Participants
  Day 3 post-administration of AP1903: complete response | 0 | 1
  Day 3 post-administration of AP1903: partial response | 0 | 0
  Day 3 post-administration of AP1903: no response | 0 | 0
  Day 3 post-administration of AP1903: progression | 0 | 0
  Day 7 post-administration of AP1903: complete response | 0 | 1
  Day 7 post-administration of AP1903: partial response | 0 | 0
  Day 7 post-administration of AP1903: no response | 0 | 0
  Day 7 post-administration of AP1903: progression | 0 | 0
  Day 14 post-administration of AP1903: complete response | 0 | 1
  Day 14 post-administration of AP1903: partial response | 0 | 0
  Day 14 post-administration of AP1903: no response | 0 | 0
  Day 14 post-administration of AP1903: progression | 0 | 0
  Day 28 post-administration of AP1903: complete response | 0 | 1
  Day 28 post-administration of AP1903: partial response | 0 | 0
  Day 28 post-administration of AP1903: no response | 0 | 0
  Day 28 post-administration of AP1903: progression | 0 | 0
  Day 56 post-administration of AP1903: complete response | 0 | 0
  Day 56 post-administration of AP1903: partial response | 0 | 0
  Day 56 post-administration of AP1903: no response | 0 | 0
  Day 56 post-administration of AP1903: progression | 0 | 1

6. Secondary Outcome: To Assess the Incidence of GvHD Treatment Failure Post-administration of AP1903.
Description: To assess the incidence of GvHD treatment failure, defined as no response, progression, administration of additional therapy for GvHD, or mortality post-administration of AP1903.
Time Frame: Day 3, 7, 14, 28, and 56 post-administration of AP1903.
Population: Patient who received AP1903
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 1
Participants
  Day 3 post-administration of AP1903. | 0 | 1
  Day 7 post-administration of AP1903. | 0 | 1
  Day 14 post-administration of AP1903. | 0 | 1
  Day 28 post-administration of AP1903. | 0 | 1
  Day 56 post-administration of AP1903. | 0 | 1

7. Secondary Outcome: To Assess the Incidence of Acute GvHD Flare After CR/PR Requiring Additional Agent for Systemic Therapy Before Day 56 Post-administration of AP1903.
Description: To assess participants with incidence of acute GvHD flare after CR/PR requiring additional agent (including 2.5 mg/kg/day of prednisone [or methylprednisolone equivalent of 2 mg/kg/day]) for systemic therapy before Day 56 post-administration of AP1903."
Time Frame: before Day 56 post AP1903
Population: Patients who received AP1903
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

8. Secondary Outcome: To Assess Post Donor Lymphocyte Infusion (DLI) Chimerism
Description: To assess the number of Participants with 100% donor chimerism at 6 months post donor lymphocyte infusion (DLI)
Time Frame: 6 months
Population: patients who received DLI
Measure: Count of Participants; unit: Participants
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 1
Participants | 0 | 1

9. Other Pre Specified Outcome: To Assess Presence of Gvhd Post Donor Lymphocyte Infusion (DLI)
Description: To assess at 6 months post donor lymphocyte infusion (DLI): GVHD grade & time to resolution
Time Frame: 6 months
Population: Patient who received DLI was removed from study prior to 6 month time frame. No outcome measure was provided.
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: To Determine the Change in Patient-reported Outcomes
Description: To determine the change in patient-reported outcomes from enrollment to day 56 post administration of AP1903, through the patient quality of life survey.
Time Frame: Day 56 post administration of AP1903
Population: Participant completed quality of life surveys but data was not analyzed to provide outcome measure.
Arm/Group | Transplant Only | Transplat Plus DLI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 30 days after DLI or after AP1903 infusion, whichever is later
Description: Adverse events were captured for patients who received DLI and AP1903.
Arm/Group | Transplant Only | Transplat Plus DLI
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transplant Only (N=0) | Transplat Plus DLI (N=1)
Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Transplant Only (N=0) | Transplat Plus DLI (N=1)
Elevated creatinine (Renal and urinary disorders) | 0 | 1
Infection (CMV) (Infections and infestations) | 0 | 1
Infection (adenovirus) (Infections and infestations) | 0 | 1
Infection (E.Coli) (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Skin Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT01875237/Prot_SAP_000.pdf